CLINICAL TRIAL: NCT03562143
Title: Daily vs Alternate Day Iron Supplementation for Pregnant Women With Iron Deficiency Anemia: A Randomized Controlled
Brief Title: Daily vs Alternate Day Iron Supplementation for Pregnant Women With Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1781
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron; Deficiency; Anemia; Supplementation; Pregnancy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Patients that agree to participate will be randomized to receive either 1 tablet of 325mg ferrous sulfate (65 mg of elemental iron) on consecutive days for 6 weeks or 2 tablets together (130 mg of elemental iron ) every other day for 6 weeks. Both groups will be receiving the same total amount of iron over the study period (2730 mg of elemental iron over 6 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate-day iron supplementation (Experimental): Patients taking iron supplementation given as 2 tabs of 325 mg ferrous sulfate (equivalent to 130 mg of elemental iron) for 6 weeks.
  Interventions: Dietary Supplement: Ferrous Sulfate
- Daily iron supplementation (Active Comparator): Patients taking iron supplementation given as 1 tab of 325 mg ferrous sulfate (equivalent to 65 mg of elemental iron) for 6 weeks.
  Interventions: Dietary Supplement: Ferrous Sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — Patients will take iron supplementation given as 2 tabs of 325 mg ferrous sulfate (equivalent to 130 mg of elemental iron) on alternate day for 6 weeks.
  Other Names: Alternate-day iron supplementation
  Arms: Alternate-day iron supplementation
Dietary Supplement: Ferrous Sulfate — Patients will take iron supplementation given as 1 tab of 325 mg ferrous sulfate (equivalent to 65 mg of elemental iron) daily for 6 weeks.
  Other Names: Daily iron supplementation
  Arms: Daily iron supplementation

SUMMARY:
Iron deficiency is thought to be the most common nutrient deficiency among pregnant women and the most common cause of anemia in pregnancy. The consequences of iron deficiency anemia are serious and can include diminished intellectual and productive capacity and possibly increased susceptibility to infection in mothers and infants, low birthweight, and premature births, hence the importance of appropriate treatment during pregnancy.

Most guidelines recommend an increase in iron consumption by about 15-30 mg/day, an amount readily met by most prenatal vitamin formulations. This is adequate supplementation for non-anemic and non-iron-deficient women. However, women with iron deficiency anemia should receive an additional 30-20 mg/day until the anemia is corrected.

It is not clear whether intermittent administration of oral iron is equivalent to once daily to rise the hemoglobin levels in pregnant women with iron deficiency anemia. Alternate day treatment with supplemental iron has been suggested as a way to improve its absorption because daily doses may suppress the mucosal uptake of iron even in the presence of iron deficiency until the intestinal mucosa completes its turnover.

Another possible factor associated with the frequency of iron dosing is related to hepcidin, the central regulatory molecule in the metabolism of iron in mammals. The synthesis of hepcidin is controlled by 3 kinds of signals: inflammation; the need for increased erythropoiesis, and an iron status signal based on plasma iron levels and iron stores. If plasma iron levels or iron stores are increased, the resulting signal increases hepcidin levels, thereby blocking iron absorption and its release from stores (liver, macrophages) and preventing iron overload.This hepcidin effect, suppressing iron absorption, could last as long as 48h.

In this study, the researchers aim to determine if alternate day dosing of iron in pregnant women with iron deficiency anemia results in improved levels of hemoglobin or hematocrit and ferritin.

Hepcidin levels will be compared between patients on daily iron supplementation versus alternate day supplementation.

The researchers will also evaluate if alternate day dosing of iron supplementation results in a better side effect profile, and with better patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with iron deficiency anemia, defined as Hb less than 11.0 or hematocrit less than 33% with ferritin 25 ug/L
* Age 18-64 years old.
* Gestational age between 12 0/7 weeks and 34 0/7 weeks.
* No other known causes of anemia (Folate or vit b12 deficiency anemia, sideroblastic anemia, thalassemia, sickle cell anemia, aplastic anemia, hemolytic anemia, anemia of chronic disease). Anemic patients with a low ferritin level and a mean corpuscular volume (MCV) >95 will have folate and vitamin B12 measured since some patients might have combined causes of anemia and might not respond as expected to iron supplementation only.

Patients will also be required to have a normal HB electrophoresis; this is a routine test obtained on all prenatal patients.

Exclusion Criteria:

* Patients currently receiving iron supplementation
* Malabsorptive and restrictive bariatric surgery
* Inflammatory bowel disease
* Irritable bowel syndrome
* Celiac disease/atrophic gastritis/Helicobacter pylori
* Active infection (ferritin can be falsely elevated since apoferritin is an acute-phase protein like CRP and increases both during infections and inflammatory reactions eg postoperatively).
* Patients with contraindications to iron supplementation such as iron overload or hypersensitivity

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 88 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin Level | baseline and 6 weeks
  The change in the level of hemoglobin in pregnant patients with iron deficiency anemia after 6 weeks of treatment with either daily or alternate-day iron supplementation.

SECONDARY OUTCOMES:
Change in Ferritin Level | baseline and 6 weeks
  Change in the level of ferritin in pregnant patients with iron deficiency anemia after 6 weeks of treatment with either daily or alternate-day iron supplementation.
Change in Fasting Hepcidin Level | Baseline and Day 43 post treatment
  At the end of the 6 weeks of treatment, hepcidin levels will be obtained on day 43 of the study. The 6-week hepcidin level will be compared to the starting hepcidin which will be drawn prior to initiating iron supplementation.
Side effects from Iron Supplementation Questionnaire | 6 weeks
  Patients will be asked to fill a questionnaire after 6 weeks to assess for adverse symptoms associated with consumption of iron including constipation, nausea, vomiting, diarrhea, abdominal pain, and headache. Each of these items is scaled from 0 (not al all) to 10 (very much), with total scale from 0-60, with higher score indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa T Chu Lam, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sloan NL, Jordan E, Winikoff B. Effects of iron supplementation on maternal hematologic status in pregnancy. Am J Public Health. 2002 Feb;92(2):288-93. doi: 10.2105/ajph.92.2.288. PMID 11818308
- [Background] Alleyne M, Horne MK, Miller JL. Individualized treatment for iron-deficiency anemia in adults. Am J Med. 2008 Nov;121(11):943-8. doi: 10.1016/j.amjmed.2008.07.012. PMID 18954837
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Short MW, Domagalski JE. Iron deficiency anemia: evaluation and management. Am Fam Physician. 2013 Jan 15;87(2):98-104. PMID 23317073
- [Background] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639
- [Background] Auerbach M, Adamson JW. How we diagnose and treat iron deficiency anemia. Am J Hematol. 2016 Jan;91(1):31-8. doi: 10.1002/ajh.24201. Epub 2015 Nov 17. PMID 26408108
- [Background] Allen LH. Anemia and iron deficiency: effects on pregnancy outcome. Am J Clin Nutr. 2000 May;71(5 Suppl):1280S-4S. doi: 10.1093/ajcn/71.5.1280s. PMID 10799402
- [Background] Breymann C. Iron Deficiency Anemia in Pregnancy. Semin Hematol. 2015 Oct;52(4):339-47. doi: 10.1053/j.seminhematol.2015.07.003. Epub 2015 Jul 10. PMID 26404445